CLINICAL TRIAL: NCT04611867
Title: Study of Supportive Application with Integrated Patient-Reported Outcomes in Patients with Advanced Pancreatic or BiliaryTract Cancer (BetterEveryDay)
Brief Title: Study of PRO in Patients with Advanced Pancreatic or Biliary Tract Cancer (BetterEveryDay)
Acronym: BetterEveryDay
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inna Chen, MD (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Inna Chen, MD, MD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AA2058
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer; Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): The intervention will be comprised of providing patients with supportive application with integrated PRO consisting of:
  * Weekly self-reporting of PRO-CTCAE with integrated preparation questionnaire available for staff
  * Daily monitoring of self-reporting by study staff
  * Intervention if required based on self-reporting
  * Reports to oncologists (at consultation)
  * Information module about treatment, side effects and contact information
  Interventions: Other: Supportive application with integrated weekly PRO
- Standard Arm (No Intervention): Standard care for patients will be included in no-intervention arm will consist of the standard procedures at Herlev Hospital, Department of Oncology for monitoring and documenting symptoms, which will be typical of oncology practice. Symptoms will be discussed and documented in the medical record during clinical encounters between patients and their oncologists. Patients will be encouraged to initiate telephone contact between visits for concerning symptoms, i.e. "call early and often".

INTERVENTIONS:
Other: Supportive application with integrated weekly PRO — Patients will fill in a web-based application PRO-CTCAE with integrated preparation questionnaire every week. If their weekly reported symptoms exceed a predefined threshold of severity, this results in a notification on the staff application interface and a nurse will contact a patient for verification of symptoms. Nurse will review patient recent treatment and PRO reports and advise patient according to the local practice for symptom management and reinforce reporting. Nurse will consult with or refers to (if possible) treating physician if patient will require medical intervention and/or physician assistance.
  Arms: Intervention Arm

SUMMARY:
Pancreatic and biliary tract cancer are ones of the leading causes of cancer-related deaths. During the course of illness, these patients often experience marked physical suffering, psychological distress and frequent unplanned resource-demanding hospitalized care. Patients with pancreatic and lung cancer have highest rates of unplanned hospitalizations. Investigator initiated prospective "Study of Supportive Application with Integrated Patient-Reported Outcomes in Patients with Advanced Pancreatic or Biliary Tract Cancer (BetterEveryDay)" is to be initiated based on the great need for optimizing treatment care, reducing hospitalizations and improving outcomes.

DETAILED DESCRIPTION:
The trial is designed as an investigator initiated prospective study of patients with advanced pancreatic or biliary tract cancer initiating systemic treatment to determine the feasibility and efficacy of supportive application with integrated weekly Patient-Reported Outcomes (PRO) on unplanned hospitalization, Quality of Life (QoL), survival, satisfaction with oncologist communication, and resource utilization.

This study will consist of Part A (Feasibility), as well as a possible Part B (Randomized controlled trial, RCT).

Initially, 30 patients with advanced lung (NSCLC) and pancreatic cancer initiating systemic therapy will be enrolled in the Part A to assess the feasibility of the supportive application with integrated weekly PRO. Patients included in feasibility Part A will be instructed in self-reporting via web-based supportive application with integrated weekly PRO.

In case of successfully completed Part A, the randomized Part B will be activated to determine the efficacy of the supportive application with integrated weekly PRO on unplanned hospitalization, QoL, survival, satisfaction and resource utilization for patients with advanced lung (NSCLC) and pancreatic cancer initiating systemic therapy. Format of that Part B will be adjusted if indicated based on the feasibility responses seen in the 30 patients in Part A. Patients will be randomized in Part B with a 1:1 ratio in a stratified manner according to cancer type (biliary tract cancer versus pancreatic cancer). If initiated, the data from Part B: RCT will be analyzed separately and will not be pooled with Part A for the purpose of statistical analysis.

Over the course of the study patients in both arms will be asked to complete questionnaires about QoL at baseline and week 12 and 24. Additionally, patients in both arms are asked to complete the modified Health Care Climate Questionnaire (HCCQ) at week 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 and over)
* Confirmed by cytology or histology advanced lung (NSCLC) or pancreatic cancer
* Written informed consent before any study procedures
* Planning to receive 1st line systemic anticancer therapy within ≤2 weeks
* Performance status: ECOG 0-2
* Access to the internet
* Ability to read and respond to questions or able to complete questions with minimal assistance required from an interpreter or family member

Exclusion Criteria:

* No mobile device
* Exhibiting signs of overt psychopathology or cognitive dysfunction
* Any medical condition that the Investigator considers significant to compromise the safety of the patient or that impairs the interpretation of study assessments
* Patient participating in another interventional study during the surveillance period. This is only relevant for studies that might interfere with the intervention. Participation in protocols related only to treatment will not preclude participation in the present study. Cases of doubt will be settled by the protocol responsible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility (Part A) | 3 months
  - Proportion of enrolled patients responding to at least two consecutive questionnaires by 12 weeks
Hospitalization (Part B) | 6 months
  - Hospitalization with any unplanned admission to the hospital and/or emergency department within the 24 weeks beginning from the day of randomization.

SECONDARY OUTCOMES:
EORTC QLQ-C30 global health status/QoL scale | 6 months
  - Adjusted mean change from baseline in global health status/QoL score from the EORTC QLQ-C30 questionnaire at 12 and 24 weeks
EORTC QLQ-C30 functional scales and symptom scales/items | 6 months
  - Adjusted mean change from baseline in functional and symptom scales from the EORTC QLQ-C30 questionnaire at 6, 12 and 24 weeks.
Overall survival | 1 year
  - Overall survival
Satisfaction with oncologist communication at 12 and 24 weeks as measured by the modified Health Care Climate Questionnaire (HCCQ) | 6 months
  - Adjusted mean in score from the modified HCCQ at 12 and 24 weeks.

OTHER OUTCOMES:
Out-of-patient care and resource utilization | 6 months
  - Time to first ER visit and/or hospitalization
Out-of-patient care and resource utilization | 6 months
  - Rates of hospital admissions
Out-of-patient care and resource utilization | 6 months
  - Mean length of hospital stay
Out-of-patient care and resource utilization | 6 months
  - Number of additional/unplanned nursing calls
Out-of-patient care and resource utilization | 6 months
  - Number of additional/unplanned out-patient care visits
Tolerability of systemic therapy | 6 months
  - Time receiving active cancer treatment

CONTACTS AND LOCATIONS:
Overall Officials: Inna M Chen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark